CLINICAL TRIAL: NCT03483506
Title: A Phase I, Open-label, Single-arm Multiple Dose Trial to Investigate Pharmacokinetics and Absolute Bioavailability of BI 1467335 Administered as an Oral Dose Simultaneously With an Intravenous Microtracer Dose of [C-14] BI 1467335 After Single and Multiple Oral Doses in Healthy Male Volunteers
Brief Title: This Study in Healthy Men Tests How the Body Takes up BI 1467335
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1386-0019; 2017-003853-41 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Drug: BI 1467335; Drug: BI 1467335 (C-14) intravenous solution

INTERVENTIONS:
Drug: BI 1467335 — Film-coated tablet
Drug: BI 1467335 (C-14) intravenous solution — Intravenous solution

SUMMARY:
The primary objective of this trial is to investigate the absolute bioavailability of BI 1467335 with an intravenous microdose formulation containing labelled [C-14] BI 1467335 and an unlabelled oral tablet formulation of BI 1467335 in healthy male subjects.

The secondary objective is the evaluation of additional pharmacokinetic parameters following the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men) study drug via seminal fluid Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Clinically significant gastrointestinal, hepatic, renal, respiratory (including but not limited to interstitial lung disease), cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Within 30 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 5 cigarettes or 1 cigar or 1 pipe per day)
* Inability to refrain from smoking on specified trial days
* Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)e the reference range that the investigator considers to be of clinical relevance
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTcF intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

- Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column) in the period of 1 year prior to screening

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, non-randomized, single arm, multiple dose design trial in healthy male participants received unlabelled oral doses of BI 1467335 (Test product 1 (T1), film coated tablet) for 28 days and in addition microtracer-radiolabelled BI 1467335 as intravenous (iv) infusions on Days 1 and 28 (Test product 2 (T2)).
Pre-assignment Details: All participants were screened for eligibility to participate in the study. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered to trial if any one of the specific entry criteria were not met.
Groups:
- BI 1467335: All participants were orally administered treatment T1 consisted of 10 milligram (mg) (2x5) film-coated tablets of BI 1467335 once daily for 28 days in the fasted state with about 240 milliliters (ml) of non-sparkling water. In addition subjects also received the two single 10 ml intravenous (iv) infusion comprised 50 microgram (μg) BI 1467335 free base, consisting a mixture of 41.15 μg unlabelled BI 1467335 and 8.85 μg [C-14] BI 1467335 on Day 1 and a mixture of 45 μg unlabelled BI 1467335 and 5 μg [C-14] BI 1467335 free base on Day 28. The infusion started 1 hour after the intake of the BI 1467335 film-coated tablets on Day 1 and Day 28 and ended 15 minutes later.
Period: Overall Study
Arm/Group | BI 1467335
Started (Started are treated) | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All subjects who received at least one dose of the trial medication.
Arm/Group | BI 1467335
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: After the First Dose: Area Under the Concentration-time Curve of BI 1467335 Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) of BI 1467335 (After Oral Administration) and [C-14] BI 1467335 (After iv Administration) on Day 1
Description: After the first dose: Area under the concentration-time curve of BI 1467335 over the time interval from 0 extrapolated to infinity (AUC0-infinity) of BI 1467335 (after oral administration) and [C-14] BI 1467335 (after iv administration) on Day 1 is presented.
  Standard Error is actually a geometric standard Error in method of dispersion. Pharmacokinetic samples were collected on Day 1 for both groups.
Time Frame: Within 2 hours (h) before and 0.25, 0.5, 0.75, 1.083, 1.417, 2, 3, 4, 6 and 8 h after BI intake. Within 2h before and 1.083, 1.25, 1.417, 1.583, 1.75, 2, 2.25, 2.75, 3.25, 3.75, 4.25, 4.75, 5.25, 6.25, 7.25, 8.25, 9.25 and 13 h after [C-14] BI intake.
Population: Pharmacokinetic (PK) set (PKS): All subjects in the TS who provided at least one primary PK parameter not excluded due to a protocol violation relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Standard Error); unit: millimole * hour/ Liter/ kilogram
Groups:
- BI 1467335 Tab: Participant were administered 2 film-coated tablets of 5 mg (2*5 mg) of BI 1467335 orally for 28 days (Day 1 to 28).
- BI 1467335 (C-14) iv: Participant were administered BI 1467335 mixed with BI 1467335 (C-14) intravenously (50 μg BI 1467335 (C-14) in 10 mL saline) as two single iv infusions (Day 1 and Day 28, infused over 15 min, 1 hour after the oral dose.
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
millimole * hour/ Liter/ kilogram | 0.35 (1.25) | 4.16 (1.25)
Statistical Analysis 1: Comparison: BI 1467335 Tab vs BI 1467335 (C-14) iv; The statistical model used for the analysis of the primary PK endpoints was an ANOVA (analysis of variance) model on the logarithmic scale. The model included effects accounting for 'subject' and 'formulation' as sources of variation; 'subject' was considered as a random effect, whereas 'formulation' was considered as a fixed effect; Test type: Other; ANOVA; Geometric mean ratio = 8.34, 90% CI 2-sided [5.88 to 11.82], Standard Deviation 50.5 — Standard deviation is actually intra individual geometric coefficient of variation. "BI 1467335 tab" arm is the numerator, while "BI 1467335 (C-14) iv" arm is the denominator

2. Primary Outcome: After the First Dose: Maximum Measured Concentration of the BI 1467335 in Plasma (Cmax ) of BI 1467335 (After Oral Administration) and [C-14] BI 1467335 (After iv Administration) on Day 1
Description: After the first dose: maximum measured concentration of BI 1467335 in plasma (Cmax ) of BI 1467335 (after oral administration) and [C-14] BI 1467335 (after iv administration) on Day 1 is presented.
  Pharmacokinetic samples were collected on Day 1 for both groups.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
nanomole/Liter (nmol/L) | 2.72 (105.0) | 0.152 (87.6)

3. Primary Outcome: Area Under the Concentration-time Curve of BI 1467335 Over the Time Interval From 0 Extrapolated to Infinity After Oral Administration of BI 1467335 and After Intravenous Administration of [C-14] BI 1467335 on Day 28 (AUC 0-infinity, 28)
Description: After the multiple doses Area under the concentration-time curve of the BI 1467335 over the time interval from 0 extrapolated to 24 h after oral administration of BI 1467335 and after intravenous administration of [C-14] BI 1467335 on Day 28 (AUC 0-infinity, 28) is presented.
  Standard Error is actually a geometric standard Error in method of dispersion. Pharmacokinetic samples were collected before and after dispense of study medication on Day 28 for both groups. Please refer to time frame for further details.
Time Frame: 5 min before and 0.25, 0.5, 0.75, 1.083, 1.417, 2, 3, 4, 6, 8, 10, 12 and 24h after BI intake. Within 1.083 before and 0.083, 0.25, 0.417, 0.583, 0.75, 1, 1.25, 1.75, 2.25, 2.75, 3.25, 3.75, 4.25, 6.25, 8.25, 12 and 24, 48 and 96h after [C-14] BI intake.
Population: PKS
Measure: Geometric Mean (Standard Error); unit: millimole*hour/ Liter/ kilogram
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
millimole*hour/ Liter/ kilogram | 37.38 (1.24) | 60.16 (1.24)
Statistical Analysis 1: Comparison: BI 1467335 Tab vs BI 1467335 (C-14) iv; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Geometric mean ratio = 62.14, 90% CI 2-sided [52.08 to 74.14], Standard Deviation 24.4 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: After Multiple Doses: Maximum Measured Concentration of BI 1467335 in Plasma of BI 1467335 After Oral Administration and [C-14] BI 1467335 After Intravenous Administration on Day 28 (Cmax, 28)
Description: After multiple doses: maximum measured concentration of the analyte in plasma of BI 1467335 after oral administration and [C-14] BI 1467335 after intravenous administration on Day 28 (Cmax, 28) is presented.
  Pharmacokinetic samples were collected before and after dispense of study medication on Day 28 for both groups. Please refer to time frame for further details.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
nanomole/Liter (nmol/L) | 92.5 (42.8) | 0.290 (19.5)

5. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of BI 1467335 After Oral Administration of BI 1467335 and After Intravenous Administration of [C-14] BI 1467335 on Day 1 (Tmax)
Description: Time from dosing to the maximum measured concentration of BI 1467335 after oral administration of BI 1467335 and after intravenous administration of [C-14] BI 1467335 on Day 1 (tmax).
  Pharmacokinetic samples were collected on Day 1 for both groups.
Time Frame: as for outcome 1
Population: PKS
Measure: Median (Inter-Quartile Range); unit: Hours (h)
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
Hours (h) | 1.08 [0.750 to 1.09] | 0.250 [0.0915 to 0.250]

6. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration of BI 1467335 After Oral Administration of BI 1467335 and After Intravenous Administration of [C-14] BI 1467335 on Day 28 (Tmax,28)
Description: Time from dosing to the maximum measured concentration of BI 1467335 after oral administration of BI 1467335 and after intravenous administration of [C-14] BI 1467335 on Day 28 (tmax,28).
  Pharmacokinetic samples were collected before and after dispense of study medication on Day 28 for both groups. Please refer to time frame for further details.
Time Frame: as for outcome 3
Population: PKS
Measure: Median (Inter-Quartile Range); unit: Hours (h)
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
Hours (h) | 1.08 [1.08 to 1.42] | 0.250 [0.167 to 0.250]

7. Secondary Outcome: Observed Terminal Half-life of BI 1467335 After Oral Administration of BI 1467335 and After Intravenous Administration of [C-14] BI 1467335 on Day 1 (t1/2)
Description: Observed terminal half-life of BI 1467335 after oral administration of BI 1467335 and after intravenous administration of [C-14] BI 1467335 on Day 1 (t1/2).
  Pharmacokinetic samples were collected on Day 1 for both groups.
Time Frame: as for outcome 1
Population: PKS
Measure: Median (Inter-Quartile Range); unit: Hours (h)
Arm/Group | BI 1467335 Tab | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12 | 12
Hours (h) | 0.751 [0.614 to 0.905] | 0.341 [0.256 to 0.780]

8. Secondary Outcome: Observed Terminal Half-life of the Analyte [C-14] BI 1467335 After Intravenous Administration on Day 28 (t1/2,28)
Description: Observed terminal half-life of the analyte [C-14] BI 1467335 after intravenous administration on Day 28 (t1/2,28).
Time Frame: Within 1.083 before and 0.083, 0.25, 0.417, 0.583, 0.75, 1, 1.25, 1.75, 2.25, 2.75, 3.25, 3.75, 4.25, 6.25, 8.25, 12 and 24, 48 and 96h after [C-14] BI 1467335 intake on Day 28.
Population: PKS
Measure: Median (Inter-Quartile Range); unit: Hours (h)
Arm/Group | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12
Hours (h) | 2.43 [1.43 to 3.79]

9. Secondary Outcome: Clearance of the Analyte [C-14] BI 1467335 After Intravenous Administration on Day 1 (CL)
Description: Clearance of the analyte [C-14] BI 1467335 after intravenous administration on Day 1 (CL).
Time Frame: Pharmacokinetic samples were taken 2 h pre-dose and at 1.083, 1.25, 1.417, 1.583, 1.75, 2 2.25, 2.75, 3.25, 3.75, 4.25, 4.75, 5.25, 6.25, 7.25, 8.25, 9.25 and 13 h after last drug administration on day 1 for [C-14] BI 1467335.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millilitre/minute (mL/min)
Arm/Group | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12
millilitre/minute (mL/min) | 14300.0 (87.2)

10. Secondary Outcome: Clearance of the Analyte [C-14] BI 1467335 After Intravenous Administration on Day 28 (CL28)
Description: Clearance of the analyte [C-14] BI 1467335 after intravenous administration on Day 28 (CL28).
Time Frame: as for outcome 8
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millilitre/minute (mL/min)
Arm/Group | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12
millilitre/minute (mL/min) | 988 (66)

11. Secondary Outcome: Volume of Distribution of the Analyte [C-14] BI 1467335 After Intravenous Administration on Day 1 (Vz)
Description: Volume of distribution of the analyte [C-14] BI 1467335 after intravenous administration on Day 1 (Vz).
Time Frame: as for outcome 9
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12
Liter (L) | 554 (128)

12. Secondary Outcome: Volume of Distribution of the Analyte [C-14] BI 1467335 After Intravenous Administration on Day 28 (Vz, 28)
Description: Volume of distribution of the analyte [C-14] BI 1467335 after intravenous administration on Day 28 (Vz, 28).
Time Frame: as for outcome 8
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | BI 1467335 (C-14) iv
Number analyzed (Participants) | 12
Liter (L) | 204 (13.4)

13. Secondary Outcome: Absolute Bioavailability (Fabs) of BI 1467335 After Oral Administration on Day 1
Description: Absolute bioavailability (Fabs) of BI 1467335 after oral administration on Day 1, F (absolute bioavailability) on Day 1 determined as ratio Day 1 (AUC 0-∞/Dose)oral/ (AUC0-∞/Dose)iv·100 per subject.
Time Frame: Pharmacokinetic samples were taken 2 h pre-dose and at 0.25, 0.5, 0.75, 1.083, 1.417, 2, 3, 4, 6 and 8 h after last drug administration on day 1 for BI 1467335.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 1467335 Tab
Number analyzed (Participants) | 12
Ratio | 0.0834 (75.9)

14. Secondary Outcome: Absolute Bioavailability of BI 1467335 After Oral Administration on Day 28 (Fabs,28)
Description: Absolute bioavailability of BI 1467335 after oral administration on Day 28 (Fabs,28), F (absolute bioavailability) on Day 28 determined as ratio Day 28 (AUC 0-∞/Dose)oral/ (AUC0-∞/Dose)iv·100 per subject.
Time Frame: as for outcome 8
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 1467335 Tab
Number analyzed (Participants) | 12
Ratio | 0.621 (35.1)

ADVERSE EVENTS:
Time Frame: From first day of study drug administration until 12 days after last drug administration, up to 40 days.
Description: Treated set (TS): All subjects who received at least one dose of study drug.
Arm/Group | BI 1467335
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335 (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Catheter site pain (General disorders) | 2
Feeling hot (General disorders) | 1
Medical device site irritation (General disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Listless (Psychiatric disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03483506/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT03483506/SAP_001.pdf